CLINICAL TRIAL: NCT06574971
Title: Pre-Post Intervention Study to Investigate the Safety, Feasibility, & Efficacy of the NeurGear ZenBud System for the Treatment of Anxiety & Anxiety-Related Symptoms
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NeurGear (Industry)
Responsible Party: Principal Investigator, Izzy Kohler, Chief Science Officer, NeurGear
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1360094
Record Dates: First submitted 2024-08-26; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Anxiety Disorders
Keywords: Anxiety disorders; low intensity focused ultrasound; auricular nerve; vagus nerve
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Primary arm (Experimental): All participants in the study we receive the intervention
  Interventions: Device: Low intensity focused ultrasound using the NeurGear Zenbud

INTERVENTIONS:
Device: Low intensity focused ultrasound using the NeurGear Zenbud — The NeurGear Zenbud is a wearable earbud that delivers low intensity focused ultrasound to the auricular branch of the vagus nerve

SUMMARY:
The goal of this clinical trial is to learn if low intensity fodused ultrasound stiulation delivered to the auricular branch of the vagus nerve works to mitigate symptoms of anxiety disorder in adults. It will also learn about the safety and feasibility of low intensity focused ultrasound stimulation. The main questions it aims to answer are:

Is low intensity ultrasound applied to the auricular branch of the vagus nerve effective for reducing the symptoms of anxiety disorders?

Is low intensity ultrasound applied to the auricular branch of the vagus nerve effective for improving quality of life and sleep for individuals who suffer from anxiety disorders?

Is low intensity ultrasound applied to the auricular branch of the vagus nerve effective for reducing the symptoms of depression for individuals who suffer from anxiety disorders?

Is the Neurgear Zenbud a safe, accessible, and feasible way of treatment for individuals who suffer from anxiety disorders?

Participants will:

Use the ZenBud device, a wearable low intensity focused ultrasound delivery device, for 5 minutes a day, every day for 4 weeks

Complete a weekly Becks Anxiety Inventory, Becks, Depression Inventory, Pittsburgh Sleep Quality Index questionnaire, and PCL-5 weekly

Complete a post study survey asking questions about subjective efficacy and quality of life improvements.

ELIGIBILITY:
Inclusion Criteria:

1. Scoring ≥ 28 on the Beck's Anxiety Inventory
2. Age 18 or older.
3. Ability to independently provide informed consent.
4. Ability to comply with the daily treatment and weekly assessments
5. Ability to communicate in English.

Exclusion Criteria:

1. Scoring below the aforementioned cutoff on the BAI
2. Inability to comply with the treatment and assessment protocol
3. Age less than 18 years.
4. Inability to provide informed consent.
5. Conditions for which ultrasound is contraindicated including cancer, pacemaker, and impaired sensory sensitivity.
6. Conditions for which vagus nerve stimulation is contraindicated including history of vagotomy.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2024-10-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Becks Anxiety Inventory | From enrollment to the end of treatment at 4 weeks
  The Beck Anxiety Inventory (BAI) is a 21-question self-report inventory that measures anxiety levels in adults and adolescents. It was written by Aaron T. Beck, M.D., and R.A. Steer. The BAI is used to assess the intensity of physical and cognitive anxiety symptoms during the past week.

SECONDARY OUTCOMES:
Pittsburg Sleep Quality Index | From enrollment to the end of treatment at 4 weeks
  The Pittsburgh Sleep Quality Index (PSQI) is a 19-question questionnaire that assesses sleep quality and disturbances over a one-month period. It's designed for clinical populations and is valid and has acceptable psychometric properties when used in men and non-pregnant women in diverse global settings.
Becks Depression Inventory | From enrollment to the end of treatment at 4 weeks
  The Beck Depression Inventory (BDI) is a 21-item self-report questionnaire that assesses the level of depression in adults. The BDI measures both cognitive and physical symptoms of depression, such as sadness, pessimism, and worthlessness. It generates a single score that indicates the severity of depression as minimal, mild, moderate, or severe. The individual scale items are scored on a 4-point continuum, with a total summed score range of 0-63. Higher scores indicate greater depressive severity.
PTSD Checklist for DSM-5 | From enrollment to the end of treatment at 4 weeks
  The Post-Traumatic Stress Disorder (PTSD) Checklist for DSM-5 (PCL-5) is a 20-item self-report tool that assesses the 20 symptoms of PTSD in adults. It's designed for people who have experienced traumatic events. The PCL-5 can help with: Monitoring symptom changes during and after treatment, Screening people for PTSD, and Making provisional PTSD diagnoses

CONTACTS AND LOCATIONS:
Locations (1):
- NeurGear, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johnson RL, Wilson CG. A review of vagus nerve stimulation as a therapeutic intervention. J Inflamm Res. 2018 May 16;11:203-213. doi: 10.2147/JIR.S163248. eCollection 2018. PMID 29844694